CLINICAL TRIAL: NCT00880945
Title: Comparison of the Electromagnetic Navigation System and Rapid on Site Evaluation Versus Conventional Bronchoscopy and Rapid on Site Evaluation: Improved Yield in Small Peripheral Lung Lesions(Original Investigation)
Brief Title: Conventional Bronchoscopy Plus Rose Versus Electromagnetic Navigation (EMN) Plus Rose in Small Peripheral Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Balbo Piero, UOA pneumologia
Other Study IDs: 2010-no-emn
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Lung Cancer; Secondary Lung Cancer; Benign Lung Lesions
Keywords: FBS; coin lesions; ENB; ROSE
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 36-40 patients: patients with small peripheral lesions who need bronchoscopy for diagnostic purposes

SUMMARY:
The aim of this study is to evaluate if Electromagnetic navigation (ENB) in combination with rapid on site evaluation (ROSE) can improve diagnostic accuracy in those patients who fail to be diagnosed with conventional fluoroscopic assisted bronchoscopy (FBS) in combination with ROSE.

ELIGIBILITY:
Inclusion Criteria:

* presence of small peripheral lung lesions (< 3 cm) in patient suitable for surgical procedure

Exclusion Criteria:

* patient with metastatic disease
* patients unfit for surgical procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral lesion suitable for surgery who need preoperative diagnosis will be studied, at first, with conventional bronchoscopy under fluoroscopic guidance. In case of non diagnostic procedure they will be candidates for ENB. All the patients will be candidates to surgical procedure in case of malignant lesions.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-04 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the percentages of diagnosis that can be obtained adding ENB to conventional bronchoscopy in the same patient | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: piero em balbo, MD, Principal Investigator — UOA PNEUMOLOGIA NOVARA
Locations (1):
- azienda ospedaliera -universitaria Maggiore della carità, Novara, novara, Italy